CLINICAL TRIAL: NCT07020377
Title: The Hepato-protective Effect of Dapagliflozin in Type 2 Diabetes Mellitus Patients (T2DM) With Nonalcoholic Fatty Liver Disease (NAFLD)
Brief Title: Dapagliflozin in Nonalcoholic Fatty Liver Disease (NAFLD) and Type 2 Diabetes Mellitus Patients (T2DM).
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amira Bisher,PhD (Other)
Collaborators: Alexandria University (Other); Egyptian Liver Hospital (Other)
Responsible Party: Sponsor-Investigator, Amira Bisher,PhD, Yasmine Essam, Bachlor, Clinical pharmacy, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dapagliflozin NAFLD
Record Dates: First submitted 2024-11-07; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-11

CONDITIONS: Diabetes Mellitus; Non Alcholic Fatty Liver Disease
Keywords: Diabetes mellitus type 2; non alcoholic fatty liver disease; hepato-protective; Dapagliflozin
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Positive control (Placebo Comparator)
  Interventions: Drug: Placebo
- Dapagliflozin 10mg (Active Comparator): The group which takes the medication (dapagliflozin)
  Interventions: Drug: Dapagliflozin (DAPA)
- Negative control (Other): healthy participants without any medication
  Interventions: Other: Negative control

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — dapagliflozin 10mg tab once daily for NAFLD patient
  Arms: Dapagliflozin 10mg
Drug: Placebo — placebo
  Arms: Positive control
Other: Negative control — Baseline sample serum without either drug or placebo
  Arms: Negative control

SUMMARY:
Nonalcoholic fatty liver disease (NAFLD) encompasses conditions such as nonalcoholic steatohepatitis (NASH), which involves liver inflammation and fibrosis resulting from steatosis, potentially leading to cirrhosis and hepatocellular carcinoma. NAFLD is intricately linked to metabolic syndrome, with insulin resistance and hyperinsulinemia as key underlying factors. particularly among individuals with type2 diabetes. NAFLD is an independent risk factor for cardiovascular events, negatively impacting life expectancy in diabetic patients, and it exacerbates insulin resistance and glucose intolerance.

Early intervention in diabetes complicated by NAFLD is vital due to associations with hepatocarcinogenesis and macrovascular complications. Sodium-glucose cotransporter2 (SGLT2) inhibitors, which promote glucose excretion and reduce insulin dependence, have shown significant hypoglycemic effects, weight reduction, and potential benefits on liver function. Dapagliflozin, a specific SGLT2 inhibitor, has been proven effective in lowering hyperglycemia in type 2 diabetes and mitigating NAFLD-related complications in animal models. This study aimed to evaluate the impact of dapagliflozin on liver function in NAFLD patients with type2 diabetes. Eligible participants received dapagliflozin for 24weeks, with assessments including body composition, serum biochemistry, and molecular parameters to determine therapeutic outcomes.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is a general term that includes nonalcoholic steatohepatitis (NASH), which is inflammation and fibrosis that accompany steatosis and can lead to hepatic cirrhosis and hepatocellular carcinoma, as well as nonalcoholic fatty liver, which is steatosis affecting hepatocytes. including diseases including diabetes, dyslipidemia, hypertension, and poor glucose tolerance, NAFLD is closely linked to metabolic syndrome due to underlying insulin resistance and related hyperinsulinemia. Thus, NAFLD can be thought of as the metabolic syndrome's hepatic manifestation. Furthermore, between 30 and 70 percent of Egyptians have NAFLD, a consequence of type 2 diabetes. NAFLD has been demonstrated to be an independent risk factor for cardiovascular events that are directly linked to the life expectancies of diabetic patients. It also aggravates insulin resistance and plays a significant role in the decline of glucose tolerance. It is crucial to carry out early and suitable therapeutic interventions for type 2 diabetes complicated by NAFLD because disorders encompassing NAFLD/NASH are closely linked to hepatocarcinogenesis and macrovascular events, which lower life expectancy in patients with diabetes. Oral hypoglycemic medications known as sodium-glucose cotransporter 2 (SGLT2) inhibitors work in a unique way by increasing the excretion of glucose in the urine and blocking the reabsorption of glucose in the proximal renal tubule. This lowers blood sugar levels without the need for insulin. SGLT2 inhibitors not only have a great hypoglycemic impact but also lower body weight and blood glucose. Additionally, they have allegedly demonstrated positive benefits on hepatic dysfunction in both clinical trials and animal models, as well as pleiotropic effects on a variety of problems and regulatory effects on macrovascular events. Therefore, when utilized to treat patients with type 2 diabetes aggravated by NAFLD, SGLT2 inhibitors should show efficacy. It has been demonstrated that dapagliflozin, a strong and specific SGLT2 inhibitor, lowers hyperglycemia in T2DM patients. In rat models, dapagliflozin has also been shown to lessen some of the problems related to NAFLD. Thus, in this study, we assessed how dapagliflozin affected the liver function of NAFLD patients with type 2 diabetes. Dapagliflozin was given to eligible individuals for 24 weeks, and body composition tests, serum biochemistry measurements, and molecular parameters were used to assess the medication's therapeutic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes mellitus patients.
* Patients were having fatty liver changes by fibro scan and with mild to moderate elevation of serum liver enzymes or without.
* patients taking insulin or anti-diabetic medications.
* Patients have Renal dysfunction.
* Patients have Cardiac problem

Exclusion Criteria:

* Patients with a history of alcohol, smoking, uncontrolled diabetes.
* Pregnancy.
* Lactation.
* Chronic liver and decompensated liver disease in hepatitis B and C.
* patients whose abdominal ultrasounds findings were extremely abnormal (mass, fibrosis, ascites, and cirrhosis) and amino transaminase levels were severely high (ALT and AST greater than 15 times the upper limit of normal according to Johns Hopkins Diabetes Guide) suggest severe liver cell injury was also worked for acute viral hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Fibroscan | 6 months
  Decrease in liver stiffness by measure CAP
soluble vascular cell adhesion molecule-1 (Svcam-1) | 6 months
  VCAM-1 was analyzed in serum using the human VCAM-1 ELISA kits.
adiponectin | 6 months
  adiponectin by enzyme-linked immunosorbent assay (ELISA).
leptin | 6 months
  leptin by enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
liver enzymes | 6 months
  ALT (alanine transaminase) and AST (aspartate transaminase)
Lipid profile | 6 months
  Cholesterol, High-density lipoprotein (HDL), Low-density lipoprotein (LDL), Triglycerides

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Egyptian liver hospital, Al Mansurah
  - Alexandria university main hospital, Alexandria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bailey CJ, Gross JL, Pieters A, Bastien A, List JF. Effect of dapagliflozin in patients with type 2 diabetes who have inadequate glycaemic control with metformin: a randomised, double-blind, placebo-controlled trial. Lancet. 2010 Jun 26;375(9733):2223-33. doi: 10.1016/S0140-6736(10)60407-2. PMID 20609968
- [Background] Wu JH, Foote C, Blomster J, Toyama T, Perkovic V, Sundstrom J, Neal B. Effects of sodium-glucose cotransporter-2 inhibitors on cardiovascular events, death, and major safety outcomes in adults with type 2 diabetes: a systematic review and meta-analysis. Lancet Diabetes Endocrinol. 2016 May;4(5):411-9. doi: 10.1016/S2213-8587(16)00052-8. Epub 2016 Mar 18. PMID 27009625
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Targher G, Day CP, Bonora E. Risk of cardiovascular disease in patients with nonalcoholic fatty liver disease. N Engl J Med. 2010 Sep 30;363(14):1341-50. doi: 10.1056/NEJMra0912063. No abstract available. PMID 20879883
- [Background] Tomah S, Hamdy O, Abuelmagd MM, Hassan AH, Alkhouri N, Al-Badri MR, Gardner H, Eldib AH, Eid EA. Prevalence of and risk factors for non-alcoholic fatty liver disease (NAFLD) and fibrosis among young adults in Egypt. BMJ Open Gastroenterol. 2021 Oct;8(1):e000780. doi: 10.1136/bmjgast-2021-000780. PMID 34610926
- [Background] Lomonaco R, Ortiz-Lopez C, Orsak B, Finch J, Webb A, Bril F, Louden C, Tio F, Cusi K. Role of ethnicity in overweight and obese patients with nonalcoholic steatohepatitis. Hepatology. 2011 Sep 2;54(3):837-45. doi: 10.1002/hep.24483. Epub 2011 Aug 8. PMID 21674556
- [Background] Browning JD, Szczepaniak LS, Dobbins R, Nuremberg P, Horton JD, Cohen JC, Grundy SM, Hobbs HH. Prevalence of hepatic steatosis in an urban population in the United States: impact of ethnicity. Hepatology. 2004 Dec;40(6):1387-95. doi: 10.1002/hep.20466. PMID 15565570